CLINICAL TRIAL: NCT06934408
Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single and Multiple Injections of HRS-5817 Injection in Healthy Adult Volunteers With or Without Obesity
Brief Title: A Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HRS-5817 Injection
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fujian Shengdi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HRS-5817-101
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Obesity; Overweight
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRS-5817 Injection Group (Experimental)
  Interventions: Drug: HRS-5817 Injection
- HRS-5817 Injection Placebo Group (Placebo Comparator)
  Interventions: Drug: HRS-5817 Injection Placebo

INTERVENTIONS:
Drug: HRS-5817 Injection — HRS-5817 injection administered subcutaneously (SC).
  Arms: HRS-5817 Injection Group
Drug: HRS-5817 Injection Placebo — HRS-5817 injection placebo administered subcutaneously (SC).
  Arms: HRS-5817 Injection Placebo Group

SUMMARY:
The purpose of this study is to assess the safety, tolerability, pharmacokinetics and pharmacodynamics of HRS-5817 when administered subcutaneously (SC) as single and multiple doses in adults who are affected by obesity.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form prior to any study-related activities, understand the procedures and methods of the study, and agree to complete this study in strict accordance with the clinical study protocol.
2. Males or females aged 18-55 years old (inclusive).
3. Subjects who are generally healthy as judged by the investigator based on medical history, vital signs, physical examination, laboratory tests and electrocardiogram (ECG) results.
4. Body weight change (difference between the maximum body weight and the minimum body weight within 3 months) of no more than 5 kg within the past 3 months.
5. Female subjects of childbearing potential must agree to take highly effective contraceptive measures and avoid egg donation from the signing of the informed consent form to 6 months after the last dose, and must have a negative blood pregnancy test result before administration and not be breastfeeding. Male subjects whose partners are women of childbearing potential must agree to take highly effective contraceptive measures and avoid sperm donation from the signing of the informed consent form to 6 months after the last dose.

Exclusion Criteria:

1. Known or suspected allergy to any ingredient in the investigational medicinal products or related products; or history of multiple and/or severe allergies to drugs or food, or history of severe anaphylaxis.
2. History of or suffering from major diseases of cardiovascular, endocrine (except primary obesity), mental, neurological, digestive, respiratory, blood, immune or genitourinary systems, which are not suitable for participation in this study as judged by the investigator.
3. Subjects who have had severe trauma or undergone major surgical procedures within 6 months before screening, or who plan to undergo surgery during the study.
4. Subjects who have participated in and used any other clinical trial drugs or medical device treatments within 3 months prior to screening or plan to do so during the study period, or within 5 half-lives of the investigational drug before screening (whichever is longer).
5. Significant changes in diet and exercise habits within 1 month before screening, or failure to maintain a basically stable lifestyle such as diet and exercise during the study.
6. Known or suspected history of drug abuse or substance abuse, or positive urine drug screening during the screening period.
7. Other situations that may interfere with the evaluation of the study results or are not suitable for participating in this study as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-05-08 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs) | Baseline up to Day 253.

SECONDARY OUTCOMES:
Area Under the curve from time 0 to time t (AUC0-t) | 0 to anticipated 253 days.
Area Under the curve from time 0 to infinity (AUC0-∞) | 0 to anticipated 253 days.
Maximum concentration (Cmax) | 0 to anticipated 253 days.
Time to reach maximum concentration (Tmax) | 0 to anticipated 253 days.
Half-life (t1/2) | 0 to anticipated 253 days.
Apparent clearance (CL/F) | 0 to anticipated 253 days.
Proportion of anti-drug antibodies (ADA) positive subjects | 0 to anticipated 253 days.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Hospital of Anhui Medical Uniersity, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided